CLINICAL TRIAL: NCT04883892
Title: BMAC vs HA in Infiltrative Therapy for Osteoarthritis of the Ankle: Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Single Injection of BMAC vs HA in the Treatment of the Ankle Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues related to the adaptation of BMAC kits to the MDR
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BMAC
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Ankle Osteoarthritis
Keywords: bone marrow aspirate concentrate; hyaluronic acid; BMAC; HA; ankle; ankle injection; ankle OA

STUDY DESIGN:
Intervention Model Description: RCT, single-blind, allocation 1:1. After 12 months patients in the control group are allowed to cross-over in the treatment group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMAC injection (Experimental): Single injection of Bone Marrow Aspirate Concentrate (BMAC) into the ankle joint
  Interventions: Procedure: BMAC
- HA injections (Active Comparator): two injections of Hyaluronic Acid (HA) into the ankle joint - one injection every 15 days.
  After 12 months patients are allowed to cross-over in the BMAC arm.
  Interventions: Procedure: HA

INTERVENTIONS:
Procedure: BMAC — patients will be injected with BMAC into the ankle joint, after treatment patients will be followed up to 24 months. In particular patients will be assessed after treatment at 1, 3, 6, 12 and 24 months.
  During the injection, samples of BMAC will be collected for the characterization of the phenotype markers and clonogenic capability
  Other Names: Bone Marrow Aspirate Concentrate injection
  Arms: BMAC injection
Procedure: HA — patients will be treated with two injection of HA, one every 15 days, into the ankle joint. After treatment these patients will be followed up to 24 months. At 12 months patients can decide to cross.over in the BMAC arm treatment. After cross-over patients will be assessed for further 12 months.
  Other Names: Hyaluronic Acid injections
  Arms: HA injections

SUMMARY:
The aim of the study is to compare the efficacy of the infiltrative therapy of BMAC vs HA up to 24 months in the treatment of the ankle osteoarthritis. The efficacy will be assessed through clinical, objective and subjective evaluations. After 12 months patients in the control group can decide to cross-over in the treatment group.

DETAILED DESCRIPTION:
All the patients who meet the inclusion criteria and giving written informed consent will be randomized. We planned to enrol 120 patients.

Following the randomization, every patient will be treated with a single injection of Bone Marrow Aspirate Concentrate (BMAC) or two injections of Hyaluronic Acid (HA) in the affected ankle.

After the treatment patients will be followed up to 24 months whit clinical and radiological assessment.

After 12 months patients in the control group can decide to cross-over in the treatment group with BMAC. These patients will be followed up further 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with degenerative ankle cartilage disease;
2. Unilateral involvement on the ankle;
3. Signs and symptoms of degenerative pathology of the ankle cartilage;
4. Radiographic or MRI signs of degenerative pathology of the ankle cartilage (OA Van Dijk grade 1-3);
5. No clinically significant electrocardiographic changes (recently performed ECG).
6. Ability and consent of patients to actively participate in clinical follow-up;

Exclusion Criteria:

1. Patients unable to give consent;
2. Patients who have undergone intra-articular infiltration of another substance in the preceding 6 months;
3. Patients who have undergone ankle surgery in the preceding 12 months;
4. Patients with malignant neoplasms;
5. Patients with rheumatic diseases;
6. Patients with uncompensated diabetes;

9. Patients with uncompensated thyroid metabolic disorders; 10. Patients who abuse alcoholic beverages, drugs or medications; 11. Body Mass Index > 35;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
AOS (Ankle Osteoarthritis Scale) | Baseline, 1, 3, 6, 12, 24 months
  Evaluation of the change from baseline of the OAS score, assessing the trend of pain and function up to 24 months from the treatment

SECONDARY OUTCOMES:
AOFAS (The American Orthopedic Foot and Ankle Score) | Baseline, 1, 3, 6, 12, 24 months
  Score 0-100 made by 3 categories: Pain (0-40), Function (0-50) and Alignment (0-10).
  The best clinical and function condition is represented by a score of 100. 0 is the worst possible condition.

OTHER OUTCOMES:
VAS function (Visual Analog Score - function) | Baseline, 1, 3, 6, 12, 24 months
  the scale is to expect the patient to select the number that best describes their functional disability status, in a range of length from 0 to 10 cm. The higher the value indicated the higher the degree of disability.
VAS pain (Visual Analog Score - pain) | Baseline, 1, 3, 6, 12, 24 months
  the scale is to expect the patient to select the number that best describes their pain status, in a range of length from 0 to 10 cm. The higher the value indicated the higher the degree of disability.
EuroQol Visual Analogue Scale (EQ-VAS) | Baseline, 1, 3, 6, 12, 24 months
  0 - 100 scale where 100 is the "best possible health"and 0 is the "worst possible health"
EQ-5D (EuroQoL) Current Health Assessment | Baseline, 1, 3, 6, 12, 24 months
  Score for the assessment of the quality of life of the patient.
Patient Acceptable Symptom State (PASS) | Baseline, 1, 3, 6, 12, 24 months
  tool for assessing patient satisfaction in consideration of their current degree of pain, function and daily activity. The patient will evaluate his degree of satisfaction by answering a dichotomous closed question (yes / no).
Evaluation of the osteoarthrosis progression of the ankle joint after treatment through radiological exams | 12, 24 months
  RX and MRI will be performed at 12 and 24 month after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shapiro SA, Kazmerchak SE, Heckman MG, Zubair AC, O'Connor MI. A Prospective, Single-Blind, Placebo-Controlled Trial of Bone Marrow Aspirate Concentrate for Knee Osteoarthritis. Am J Sports Med. 2017 Jan;45(1):82-90. doi: 10.1177/0363546516662455. Epub 2016 Sep 30. PMID 27566242
- [Background] Kennedy JG, Murawski CD. The Treatment of Osteochondral Lesions of the Talus with Autologous Osteochondral Transplantation and Bone Marrow Aspirate Concentrate: Surgical Technique. Cartilage. 2011 Oct;2(4):327-36. doi: 10.1177/1947603511400726. PMID 26069591
- [Background] Giannini S, Buda R, Cavallo M, Ruffilli A, Cenacchi A, Cavallo C, Vannini F. Cartilage repair evolution in post-traumatic osteochondral lesions of the talus: from open field autologous chondrocyte to bone-marrow-derived cells transplantation. Injury. 2010 Nov;41(11):1196-203. doi: 10.1016/j.injury.2010.09.028. Epub 2010 Oct 8. PMID 20934692
- [Background] Buda R, Vannini F, Castagnini F, Cavallo M, Ruffilli A, Ramponi L, Pagliazzi G, Giannini S. Regenerative treatment in osteochondral lesions of the talus: autologous chondrocyte implantation versus one-step bone marrow derived cells transplantation. Int Orthop. 2015 May;39(5):893-900. doi: 10.1007/s00264-015-2685-y. Epub 2015 Feb 8. PMID 25662594
- [Background] Vannini F, Cavallo M, Ramponi L, Castagnini F, Massimi S, Giannini S, Buda RE. Return to Sports After Bone Marrow-Derived Cell Transplantation for Osteochondral Lesions of the Talus. Cartilage. 2017 Jan;8(1):80-87. doi: 10.1177/1947603516642574. Epub 2016 Apr 12. PMID 27994723
- [Background] Luciani D, Cadossi M, Tesei F, Chiarello E, Giannini S. Viscosupplementation for grade II osteoarthritis of the ankle: a prospective study at 18 months' follow-up. Chir Organi Mov. 2008 Dec;92(3):155-60. doi: 10.1007/s12306-008-0066-z. Epub 2008 Dec 6. PMID 19067120